CLINICAL TRIAL: NCT05588687
Title: The Effect of Two Different Distraction Methods Applied During Venous Blood Collection Procedure on the Level of Pain, Fear and Anxiety in Pediatric Emergency Department
Brief Title: The Effect of Two Distraction Methods on the Level of Pain, Fear and Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Remziye Semerci, Assistant Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Koç University
Record Dates: First submitted 2022-08-30; First posted 2022-10-20 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Pain; Anxiety; Fear; Venipuncture Site Reaction; Nursing Caries
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Intervention Model Description: This study is an experimental, parallel-group (intervention-control), randomized controlled design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Children in the control group will be received standard care. Control group children will not receive any distraction techniques.
- Virtual reality group (Experimental): The children in the VR groups will watch the video by wearing virtual glasses during the blood draw. By wearing the VR headsets in the VR-Rollercoaster Group, will watch Ice Age.
  Interventions: Behavioral: Virtual reality
- Tablet group (Experimental): The children in the tablet groups will watch the video during the blood draw with tablet. They will watch Ice Age.
  Interventions: Device: Tablet

INTERVENTIONS:
Behavioral: Virtual reality — Children will watch Ice Age in virtual reality during blood draw and the researcher will monitor their pain, anxiety and fear.
  Arms: Virtual reality group
Device: Tablet — Children will watch Ice Age with a tablet during blood draw and the researcher will monitor their pain, anxiety and fear.
  Arms: Tablet group

SUMMARY:
The aim of this study is to determine the effect of watching cartoons with virtual reality glasses and tablets applied during the blood collection process on the level of pain, fear and anxiety experienced by children.

DETAILED DESCRIPTION:
Needle procedures applied to children for diagnosis and treatment cause fear, anxiety, and pain. In cases where children's pain and fear cannot be controlled, health professionals and parents may experience feelings of stress, helplessness, and guilt. Many approaches reduce pain and anxiety in children during painful procedures. The most commonly used of these approaches is the distraction technique, also known as the distraction technique, which is constructed with cognitive and behavioral processes. There are many methods used to divert attention. Some of those; watching cartoons, inflating balloons, creating balloons by blowing foam, directing techniques, parent coaching, using virtual reality (VR) glasses, listening to music, kaleidoscope, and using distraction cards. The research is a randomized controlled experimental study designed to determine the effects of two different methods (watching 360-degree cartoons with virtual reality glasses and watching cartoons with a tablet) during the blood collection procedure in children, on the level of pain, fear, and anxiety experienced by children.

ELIGIBILITY:
Inclusion Criteria:

* The child and family agree to participate in the research,
* The child is between the ages of 5-12
* The child does not have a chronic and mental health problem.
* Not having a visual and hearing disability
* No history of sedative, analgesic or narcotic substance use within 24 hours before admission
* Not having a febrile illness at the time of application
* Absence of a disease causing chronic pain
* Being treated in the green area according to the 3-level (red-yellow-green) triage system.
* Performing the operation at once

Exclusion Criteria:

* • The child and family's refusal to participate in the research

  * Having a visual and auditory problem
  * The child is less than 5 years old or older than 12 years old
  * The child has a chronic and mental health problem
  * Being treated in the red or yellow area according to the 3-level (red-yellow-green) triage system.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Pain assesed by Wong-Baker FACES | 1 minute before the blood draw procedure
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst). This scale was assessed using self-report and reports from the parents, the researcher and the nurse who attempted the blood draw after the blood draw procedure in this study.
Pain assesed by Wong-Baker FACES | 1 minute after the blood draw procedure
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst). This scale was assessed using self-report and reports from the parents, the researcher and the nurse who attempted the blood draw after the blood draw procedure in this study.
Procedure Related Fear | 1 minute before the blood draw procedure
  The Child Fear Scale (CFS) used. This scale is a one-item self-report measure for measuring pain-related fear in children. This one-item scale consists of five sex-neutral faces. It ranges from a no fear (neutral) face on the far left to a face showing extreme fear on the far right. The rater responds indicates the level of fear. It can be used by the parents and researchers before and during the procedure for children aged 5-10 years.CFS were administered by the researcher to the children to assess their fear levels about blood draw before and after blood draw procedure.
Procedure Related Fear | 1 minute after the blood draw procedure
  The Child Fear Scale (CFS) used. This scale is a one-item self-report measure for measuring pain-related fear in children. This one-item scale consists of five sex-neutral faces. It ranges from a no fear (neutral) face on the far left to a face showing extreme fear on the far right. The rater responds indicates the level of fear. It can be used by the parents and researchers before and during the procedure for children aged 5-10 years.CFS were administered by the researcher to the children to assess their fear levels about blood draw before and after blood draw procedure.
Procedure Related Anxiety | 1 minute before the blood draw procedure
  The Children's Anxiety Meter (CAM) used. It assesses children's anxiety in clinical settings and uses before medical procedures. The CAM is drawn like a thermometer with a bulb at the bottom, also includes horizontal lines at intervals going up to the top. Children are asked to mark how he/she feel "right now" to measure state anxiety (CAM-S). (Kleiber & Mccarthy, 2006). Scores range from 0 to 10. It validated at children aged 4-10 years during an intravenous procedure.CAM were administered by the researcher to the children to assess their anxiety levels about blood draw before and after the blood draw procedure.
Procedure Related Anxiety | 1 minute after the blood draw procedure
  The Children's Anxiety Meter (CAM) used. It assesses children's anxiety in clinical settings and uses before medical procedures. The CAM is drawn like a thermometer with a bulb at the bottom, also includes horizontal lines at intervals going up to the top. Children are asked to mark how he/she feel "right now" to measure state anxiety (CAM-S). (Kleiber & Mccarthy, 2006). Scores range from 0 to 10. It validated at children aged 4-10 years during an intravenous procedure.CAM were administered by the researcher to the children to assess their anxiety levels about blood draw before and after the blood draw procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Remziye Semerci, PhD, Principal Investigator — Koç University
Locations (1):
- Remziye Semerci, Edirne, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No